CLINICAL TRIAL: NCT07228143
Title: Stepped Care Cognitive Behavioral Therapy for Children and Adolescents With Anxiety
Brief Title: Stepped Care Treatment for Anxiety Resilience
Acronym: STAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Wiese (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Andrew Wiese, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-58155
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Generalized Anxiety Disorder (GAD); Social Anxiety Disorder (SAD); Separation Anxiety Disorder; Specific Phobia; Obsessive Compulsive Disorder (OCD); Panic Disorder (With or Without Agoraphobia)
Keywords: Anxiety; Child; Adolescents; Obsessive compulsive disorder; stepped care; psychotherapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation; Phobia, Specific; Obsessive-Compulsive Disorder; Panic Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-care treatment model compared to active control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation and Mentorship Training (Active Comparator): Families randomized to Relaxation and Mentorship Training (RMT) will receive 14 sessions of relaxation training to match intervention dosage in STEP-A. RMT is a multi-component relation-based protocol for children and adolescents experiencing anxiety. Initially designed as a control condition in multiple RCTs for CAD, the protocol integrates evidence-based relaxation strategies with non-anxiety specific elements, such as autobiographical writing. Sessions 1-7 will occur weekly across seven weeks to align timing of sessions 1-4 in Step 1 of STEP-A. Aligning the timing of Sessions 1-4 allows us to test treatment mechanisms, ensures equipoise between arms for cost-effeteness analyses keeping treatment durations equivalent. To ensure children in both conditions receive a full 14-sessions of therapy the last 4 sessions of RMT are staggered to mimic the staggering of SPACE in step one.
  Interventions: Behavioral: Relaxation and Mentorship Training (RMT)
- Stepped Care Targeting Exposure and Parenting for Anxiety (STEP-A) (Experimental): STEP-A is a two-step treatment with Step 1 an abbreviated version of SPACE, which has demonstrated comparable efficacy to standard SPACE for CAD and OCD. In Step 1, parents read Breaking Free of Child Anxiety and OCD and engage in therapeutic tasks with their child while meeting with the therapist for four, 45-minute sessions at weeks 2, 4, 6, and 8. STEP-A Step 1 responders proceed to a 10-week maintenance period to practice skills learned.
  Step 2 consists of PCET, an empirically validated family-based CBT protocol designed to treat CAD more effectively and efficiently than traditional CBT by emphasizing exposures and increasing parental involvement to maximize generalization. Ten weekly sessions with the therapist. Sessions 1 and 2 include psychoeducation and development of exposure hierarchy, while sessions 3, onward, emphasize in-session exposure practice and identifying between-session exposure homework, with parents leading in-session exposures starting session 5, onward.
  Interventions: Behavioral: Stepped Care Targeting Exposure and Parenting for Anxiety (STEP-A)

INTERVENTIONS:
Behavioral: Relaxation and Mentorship Training (RMT) — RMT is a multi-component relation-based protocol for children and adolescents experiencing anxiety. Initially designed as a control condition in multiple RCTs for CAD, the protocol integrates evidence-based relaxation strategies with non-anxiety specific elements, such as autobiographical writing
  Arms: Relaxation and Mentorship Training
Behavioral: Stepped Care Targeting Exposure and Parenting for Anxiety (STEP-A) — STEP-A is a two-step treatment with Step 1 an abbreviated version of SPACE, which has demonstrated comparable efficacy to standard SPACE for CAD and OCD. In Step 1, parents read Breaking Free of Child Anxiety and OCD and engage in therapeutic tasks with their child while meeting with the therapist for four, 45-minute sessions at weeks 2, 4, 6, and 8. STEP-A Step 1 responders proceed to a 10-week maintenance period to practice skills learned.
  Step 2 consists of PCET, an empirically validated family-based CBT protocol designed to treat CAD more effectively and efficiently than traditional CBT by emphasizing exposures and increasing parental involvement to maximize generalization. Ten weekly sessions with the therapist. Sessions 1 and 2 include psychoeducation and development of exposure hierarchy, while sessions 3, onward, emphasize in-session exposure practice and identifying between-session exposure homework, with parents leading in-session exposures starting session 5, onward.
  Arms: Stepped Care Targeting Exposure and Parenting for Anxiety (STEP-A)

SUMMARY:
Childhood anxiety disorders (CAD) are common and impairing. Family based cognitive behavioral therapy (CBT) is efficacious in treating CAD. Yet, many children do not receive care due to barriers such as limited provider availably, high treatment costs, and constrained family resources (e.g., time). To combat these barriers, other treatment methods have been developed.

The stepped care treatment models maximize resources by providing low-intensity, low-cost interventions as a first time treatment, while stepping up care for those needing more intensive treatment. Specifically, a stepped care model for CAD that begins with a parent-focus intervention has great promise to deliver efficacious and cost-effective treatment without having to engage the child.

While stepped care approaches show promise in treating CAD with comparable efficacy to standard CBT, there remains a large research-to-practice gap. The stepped care model for CAD that begins with a parent-focused intervention has yet been explored, and very little is known about intervention mediators that explain mechanisms of change.

This research is being done to improve the reach and quality of services using a stepped care model, offering an affordable and practical solution to the widespread gap in youth mental health care.

DETAILED DESCRIPTION:
Anxiety disorders in children and adolescents (CAD) are common and confer significant impairment in academic, peer, and family functioning. If left inadequately treated, CAD remains chronic and increases the risk of physical and mental health problems, unemployment, substance use disorders, and suicidality in adulthood. Family-based cognitive behavioral therapy (CBT) has demonstrated efficacy in the treatment of CAD. Yet, many children do not receive care due to barriers such as limited provider availability, high treatment cost, and familial constraints (e.g., time). Effective, personalized treatment approaches that are accessible, efficient, and cost-effective are needed. To combat these barriers, other treatment methods have been developed.

A stepped care model for CAD that begins with a parent-focus intervention has great promise to deliver efficacious and cost-effective treatment without having to engage the child. Stepped care is an alternative low-intensity parent focused delivery system that incorporates the best available evidence to treat CAD within a stepped care model, which utilizes task-shifting with parent involvement, honoring the role of parents in helping their children.

*The hypothesized treatment mechanisms include parent-focused targets (i.e., family accommodation, parental distress) and child-focused targets (i.e., emotional processing, inhibitory learning) and child-focused targets (i.e., emotional processing, inhibitory learning). The stepped care model would task-shift therapeutic components to parents using scalable multi-media-based content.

Although stepped care approaches show promise in treating CAD with comparable efficacy to standard CBT, there remains a large research-to-practice gap and very little is known about intervention mediators that explain mechanisms of change.

This research is being done to understand and improve the reach and quality of services using a stepped care model, offering an affordable and practical solution to the widespread gap in youth mental health care.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of OCD or an anxiety disorder including separation anxiety disorder, social phobia, generalized anxiety disorder, specific phobia, agoraphobia, panic disorder, as determine by an IE using the DIAMOND-KID diagnostic interview.
* Score of ≥ 14 on the PARS (items 2-7) which corresponds to clinically significant anxiety.
* The child is 7-17 years old.
* Residence in Texas and located in the state of Texas during treatment sessions.

Exclusion Criteria:

* -Psychosis, cognitive disability, any condition that would limit the caregiver's ability to follow instructions.
* Parent substance use disorder within the past 3 months, which could impact their ability to implement step 1
* Child or parent is suicidal. A delayed entry once the parent or child is stabilized (>6 months post suicidality) and no longer has suicidal ideation will be allowed if appropriate.
* New pharmacological interventions or treatment changes: Initiation of an antidepressant within 12 weeks before study enrollment or 6 weeks for an antipsychotic, benzodiazepine, or attention deficit hyperactivity disorder (ADHD) medication before enrollment, or any change in established psychotropic medication (e.g., antidepressants, anxiolytics) within 6 weeks before study enrollment (4 weeks for antipsychotic, anti-anxiety, benzodiazepine, or ADHD medication changes). Medications will remain stable during treatment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale | Baseline (before treatment or week 1), midway point (week 8), stepped care treatment (7 weeks), PCET during treatment (10 weeks), post (week 20), 1 month follow-up (week 24), caregiver interview (week 32)
  The Pediatric Anxiety Rating Scale is a clinician-administered measures of pediatric anxiety symptom and symptom severity, that can be used across a broad range of anxiety-related disorders. The first part of the measure consists of a symptom checklist where responses are recorded from both the child and caregiver/parent to index the various types of anxiety the child experiences. The second part is a 7-item symptom severity scale where responses are recorded using a 0 ("no symptoms") to 5 ("extreme") Likert-type scale. Different scoring methods can be used, including a 5-item scoring (range = 0 - 25), that is preferred for clinical trial research, and is calculated using the sum of items 2, 3, 5, 6, and 7; this approach excludes items assessing overall number of anxiety symptoms and somatic symptoms. Higher scores are suggestive of more severe anxiety.
The Clinical Global Impression-Severity | Baseline (before treatment or week 1), midway point (week 8), stepped care treatment (7 weeks), PCET during treatment (10 weeks), post (week 20), 1 month follow-up (week 24), caregiver interview (week 32)
  The Clinical Global Impression-Severity is a single-item rating of symptom severity that can be used across a broad range of mental health conditions. The measure asks the rater to assess the overall severity of the individual's illness with response options ranging from 1 ("normal; no illness") to 7 ("among the most extremely ill patients").
The Clinical Global Impression-Improvement | Baseline (before treatment or week 1), midway point (week 8), stepped care treatment (7 weeks), PCET during treatment (10 weeks), post (week 20), 1 month follow-up (week 24), caregiver interview (week 32)
  The Clinical Global Impressions-Improvement Scale is a single-item assessment measure used to assess overall improvement in symptoms relative to baseline. Responses are recorded using a 1 ("very much worse) to 7 ("very much improved") scale, with the midpoint, 4, reflecting "no change" since baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be available to others outside of the study protocol due to concerns o participant confidentiality and sensitivity surrounding mental health symptoms assessed.

REFERENCES:
- [Background] Whiteside SPH, Sim LA, Morrow AS, Farah WH, Hilliker DR, Murad MH, Wang Z. A Meta-analysis to Guide the Enhancement of CBT for Childhood Anxiety: Exposure Over Anxiety Management. Clin Child Fam Psychol Rev. 2020 Mar;23(1):102-121. doi: 10.1007/s10567-019-00303-2. PMID 31628568
- [Background] Cervin M, Kendall PC, Piacentini JC, Gosch EA, Wood JJ, Schneider SC, Salloum A, Birmaher B, Guzick AG, Mataix-Cols D, Storch EA. Assessing reliable change, MCID, treatment response, and remission using the Pediatric Anxiety Rating Scale (PARS) in youth with anxiety disorders. J Anxiety Disord. 2025 Sep 11;115:103070. doi: 10.1016/j.janxdis.2025.103070. Online ahead of print. PMID 40946358
- [Background] Storch EA, Salloum A, King MA, Crawford EA, Andel R, McBride NM, Lewin AB. A RANDOMIZED CONTROLLED TRIAL IN COMMUNITY MENTAL HEALTH CENTERS OF COMPUTER-ASSISTED COGNITIVE BEHAVIORAL THERAPY VERSUS TREATMENT AS USUAL FOR CHILDREN WITH ANXIETY. Depress Anxiety. 2015 Nov;32(11):843-52. doi: 10.1002/da.22399. Epub 2015 Sep 14. PMID 26366886
- [Background] Whiteside SPH, Biggs BK, Geske JR, Gloe LM, Reneson-Feeder ST, Cunningham M, Dammann JE, Brennan E, Ong ML, Olsen MW, Hofschulte DR. Parent-coached exposure therapy versus cognitive behavior therapy for childhood anxiety disorders. J Anxiety Disord. 2024 Jun;104:102877. doi: 10.1016/j.janxdis.2024.102877. Epub 2024 May 18. PMID 38788593
- [Background] Storch EA, Guzick AG, Ayton DM, Palo AD, Kook M, Candelari AE, Maye CE, McNeel M, Trent ES, Garcia JL, Onyeka OC, Rast CE, Shimshoni Y, Lebowitz ER, Goodman WK. Randomized trial comparing standard versus light intensity parent training for anxious youth. Behav Res Ther. 2024 Feb;173:104451. doi: 10.1016/j.brat.2023.104451. Epub 2023 Dec 17. PMID 38154287